CLINICAL TRIAL: NCT03219593
Title: A Prospective Study of the Efficacy and Safety of Apatinib Monotherapy as First-Line Treatment in Elderly Patients With Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Apatinib as the First-Line Therapy in Elderly Locally Advanced or Metastatic Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Principal Investigator, Qiong Wu, Principal Investigator, The First Affiliated Hospital of Bengbu Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BYEC20170710
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Gastric Cancer; Apatinib; Biomarker
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib

STUDY DESIGN:
Intervention Model Description: Apatinib Monotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib Group (Experimental): take apatinib orally (500mg/d, once a day, continuously)
  Interventions: Drug: Apatinib mesylate tablets

INTERVENTIONS:
Drug: Apatinib mesylate tablets — Apatinib is taken 500 mg every day orally, half hour after breakfast with warm water. The drug is taken 4 weeks one cycle until disease progression or intolerable toxicity or death. The dose of the study drug may be decreased to 250 mg/d following the occurrence of a clinically significant adverse event (AE). Treatment will be discontinued if the subject is unable to tolerate a daily dose of 250 mg.

SUMMARY:
The study is to investigate the efficacy and safety of apatinib for the first-fine treatment in elderly patients with locally advanced or metastatic adenocarcinoma of stomach or gastroesophageal junction, unable or unwilling to chemotherapy, through progression-free survival (PFS). Apatinib will be given to patients with an efficacy assessment of stable disease (SD), partial response (PR), or complete response (CR) every 2 cycles. Patients were assigned to 500 mg/d apatinib continually until disease progression or intolerable toxicity or patients withdrawal of consent. The dose of apatinib may be decreased to 250 mg/d following the occurrence of a clinically significant adverse event (AE). Treatment will be discontinued if the subject is unable to tolerate a daily dose of 250 mg, and the sample size is about 30 individuals. Tumor tissue samples will be collected from each enrolled subjects before the start of treatment, and detected using next generation sequencing (NGS)-based comprehensive genomic profiling. The potential biomarkers in predicting apatinib efficacy or safety will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven primary locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma;
2. Age ≥ 65 years;
3. ECOG Performance Status: 0-2;
4. No previous anti-cancer therapy for the locally advanced or metastatic disease;
5. Unable or unwilling to chemotherapy;
6. At least one measurable lesion as defined by RECIST 1.1;
7. With acceptable hematologic, cardiac, hepatic, pulmonary and renal function;
8. Can take apatinib orally;
9. Life Expectancy: 3 months or more.

Exclusion Criteria:

1. History of other primary malignancy (except basal cell skin cancer or cervical carcinoma in situ);
2. Patients with un-controlled blood pressure on medication (> 140/90 mmHg);
3. Patients with other nonmeasurable disease such as un-controlled diabetes, severe cardiovascular and cerebrovascular diseases;
4. Patients with bleeding tendency, receiving thrombolytics or anticoagulants；
5. Patients with massive hydrothorax or ascites;
6. Patients with uncontrolled central nervous system (CNS) metastases;
7. Proteinuria 2+ or 24-hour urinary protein ≥ 1g;
8. History of drug addiction or abuse;
9. Patients cannot take apatinib orally for any reason;
10. Estimated life expectancy ˂ 3 months;
11. Current, recent (within 4 weeks prior to study entry), or planned participation in any other clinical trials;
12. Inability to understand and agree to informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-07 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 1 year
  PFS was defined to be the time from registration to the date of disease progression or death resulting from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
  OS was defined to be the time from registration to the date of death resulting from any cause or the last contact.
Disease control rate (DCR) | 1 year
  DCR was defined as the proportion of patients who achieved complete response (CR ), partial response (PR) and stable disease (SD) for at least 8 weeks.
Objective response rate (ORR) | 1 year
  ORR was defined as the proportion of eligible patients who achieved a confirmed CR or PR by RECIST 1.1 criteria evaluated by the investigators.
Quality of life score (QoL) | 1 year
  QoL is a questionnaire developed to assess the quality of life of cancer patients.
Adverse Events(AEs) | 1 year
  AEs are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v4.0.

OTHER OUTCOMES:
Tumor biomarkers | Before the start of apatinib treatment
  Tumor tissue samples will be applied to next generation sequencing (NGS) detection to reveal any gene variation through comprehensive genomic profiling.

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Wu, M.D.,Ph.D, Principal Investigator — First Affiliated Hospital of Bengbu Medical College
Locations (1):
- Department of Medical Oncology, First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No